







**FULL/LONG TITLE OF THE TRIAL:** To Co-develop and test an eHealth Intervention tO improve knowledge, attItude and experienCE in patients living with an Implantable Cardioverter Defibrillator

| Defibrillator | | |
|---|---|---|
| SHORT TRIAL TITLE / ACRONY | M: CHOICE-ICD | |
| RESEARCH REFERENCE NUMI | BERS: | |
| IRAS Number:<br>ISRCTN Number / Clinical<br>trials.gov Number: | IRAS ID 343944 | |
| SPONSORS Number: | B24/05 | |
| FUNDERS Number: | BHF Case Reference FS | /CDRF/22/21048 |
| PROTOCOL VERSION NUMBER | R AND DATE: Version 2.3 | 6 <sup>th</sup> June2024 |
| SPONSOR: Queen's University B | elfast | |
| For and on behalf of the Trial S | Sponsor: | |
| Name (please print): | | Date:// |
| Kathryn Taylor | | |
| Research Governance, Ethics & University, Belfast | Integrity, at Queen's | |
| Chief Investigator: | | |
| Signature: | | Date: |
| Name: (please print): | | |









## **LIST of CONTENTS**

| GENERAL INFORMATION | Page No. |
|---------------------------------------------------------|----------|
| TITLE PAGE | 1 |
| RESEARCH REFERENCE NUMBERS | 1 |
| SIGNATURE PAGE | 1 |
| i. LIST of CONTENTS | 2 |
| ii. FUNDING | 3 |
| iii. TRIAL FLOW CHART | 3 |
| SECTION | |
| 1: ABSTRACT | 4 |
| 2: BACKGROUND AND PILOT WORK | 4-7 |
| 3. AIM & OBJECTIVES | 7 |
| 4. TRIAL DESIGN | 8-9 |
| 5: POWER CALCULATION & PARTICIPANT ELIGIBILITY CRITERIA | 9-10 |
| 6. INTERVENTION | 10 |
| 7. DATA COLLECTION & OUTCOME MEASURES | 11 |
| 8. DATA ANALYSIS | 11-12 |
| 9. TRIAL MONITORING | 12 |
| 10. TRIAL MANAGEMENT | 12 |
| 11. ETHICS | 12 |
| 12. DISSEMINATION POLICY | 13 |
| 13. REFERENCES | 13-16 |
| 14. APPENDICES | 17 &18 |

### **FUNDING AND SUPPORT IN KIND**

| FUNDER(S) | FINANCIAL AND NON FINANCIALSUPPORT GIVEN |
|--------------------------|------------------------------------------|
| British Heart Foundation | £315,794.50 over 36 months |









## **Trial Flow Chart (Figure 1)**











## 1: Abstract

Implantable cardioverter defibrillator (ICD) is cornerstone in the treatment of life-threatening arrhythmias, yet 25% of patients report poor quality of life following implantation.

**Aim:** To co-design, optimize and establish feasibility and acceptability of eHealth intervention: CHOICE-ICD website, to reduce anxiety and improve patient involvement in future palliative decisions.

**Methods**: Phase 1: Underpinned by theory and research, core components of an intervention was co-designed according to a six-step process, in collaboration with stakeholders. Components included ICD written information, educational animations, virtual reality (VR) application, patient and care videos and a communication "prompt" for consultations. An expert advisory group oversaw the iterative development, user testing (n=10) and optimization. Phase 2: CHOICE-ICD is a prospective study, recruiting 128 patients awaiting or recently implanted ICD or cardiac resynchronisation therapy with ICD (CRTd) from Northern Ireland and Glasgow Participants will use the intervention for 3 months. Data will be analyzed to determine feasibility and acceptability.

**Outcomes:** Recruitment, consent and randomization rates, and completion of questionnaires at baseline,3 and 6 months. Acceptability of intervention delivery and suitability of outcome measures.

**Conclusions:** First UK eHealth intervention that will provide information to patients with an ICD, tailored to their needs. According to outcomes, plans will be initiated for future effectiveness trial.

## 2: Background to the project and pilot data

# Identification of the problem: Unmet psycho-educational needs

Implantable Cardioverter Defibrillators (ICDs) are recognised as an effective treatment for life-threatening arrhythmias (1), contributing to a worldwide rise in implantation rates. Within the United Kingdom (UK) over 6 thousand ICDs were implanted in 2015 (2), with Northern Ireland (NI) health service implanting a total of 156 devices per million population annually (2016/2017(3)). The combination of Cardiac Resynchronisation Therapy, which is a 3-lead









pacemaker and ICD (CRTd) has transformed heart failure treatment over the last decade, resulting in improved symptoms and quality of life, along with a reduction in hospitalisations and mortality (4, 5). Referral for implantation or battery/generator replacement remains guideline-driven (5, 6), with clinical indicators informing the decision (1, 7, 8). Clinical trials show a short-term improvement in patients' quality of life (9, 10) following ICD implantation, however for some people, the device has a detrimental impact on their psychological well-being and quality of life (11-13), particularly patients who receive frequent ICD shocks. Factors found to contribute to poor outcomes include Type D personality (14), poor illness perceptions (15), unrealistic expectations of treatment and underlying disease progression. Insufficient information can cause patients to misunderstand the functionality of their ICD, overestimating its benefits and prompting maladaptive coping strategies (16). American and Irish studies found 37% to 65% of patients with a recently implanted ICD, were unable to recall or inaccurately recalled the information professionals provided (17, 18). Similar results were noted in NI and Denmark regarding ICD deactivation (19, 20) as nearly half of patients surveyed (48%) reported they received no information. International guidelines state that providing patients with comprehensive information at the implantation stage is critical for ensuring the validity of informed consent (16, 18) as it facilitates an accurate understanding of the device capability and functionality now, and as the clinical condition progresses.

### Identifying the evidence: Interventions to inform & support patients with ICD

Effective pre-implantation education has been shown to improve knowledge, psychological acceptance and adaptation to living with the device (11, 21). International guidance recommends patients receive ongoing education and support to facilitate active involvement and improve adherence to measures for long-term health (5, 22, 23). Published guidelines provide healthcare professionals with the necessary knowledge to optimally manage patients with an ICD near the end-of-life (24, 25). Nevertheless, all too often patients reach the palliative stages, unprepared both educationally and psychologically to make informed choices concerning their device. Many professionals working across all clinical settings, in an effort to preserve the patient's hope, are reluctant to initiate a discussion about deactivation(19, 26). Deactivation is a non-invasive process, whereby the shock function of the device is 'turned off',









while remaining functions remain active. At the palliative stage of care patients and family members should be fully informed and involved in decisions concerning future treatment and care provision (27, 28).

In general, patients receive information about their device from professionals, information booklets, device manufacturer brochures or by accessing the internet (29). As a consequence of the Covid pandemic, nearly all adults in the UK now have internet access, with the proportion of those aged over 75 years increasing from 29% (2013) to 54% in 2020 (30). Technological innovation that provides personalised education and support to empower self-management has grown in acceptability with patients (31). Audio-visual aids (32) and an interest in educational virtual reality platforms are wide-reaching, sustainable and cost-effective, and can effectively provide information in a format, and at a time and place convenient to the user. Predictive modelling offered by Artificial Intelligence now makes it possible to personalise educational strategies, in accordance with, for example informational wishes, cognitive ability and clinical status of the patient (33).

A recent systematic review and meta-synthesis, on the perceptions and experiences of patients living with an ICD concluded that interventions should be patient-centric and tailored to patients' holistic needs (34). ACQUIRE-ICD, is an ongoing Danish randomised control trial (35) of a supportive intervention, incorporating cognitive behavioural therapy and psychologist input over a 12-month period. Its primary outcome is device acceptability with secondary outcomes being clinical and cost effectiveness. The CHOICE-ICD study will compliment this study, by codesigning and testing a psycho-educational intervention that integrates practical information, visual aids, patient stories and gamification. In addition to the acceptability and feasibility of the intervention, a composite outcome - knowledge, attitudes and experience, will be measured. This study has developed an intervention to provide tailored information and support, which will require wider testing to enable patients be better equipped and empowered to live well with their device. Therefore, a modern solution for what is increasingly a common clinical problem.

### Theory and pilot work: A New approach for ICD patients

Psycho-educational interventions are 'complex interventions' consisting of multiple interacting components (36). Exploratory work by this research team has identified the importance of









personalized information and support, beginning at pre-implantation and continuing throughout the illness trajectory (19, 37-39). A stakeholder meeting held in September 2021 with cardiologists, electro-physiologists, nurses, software developers, researchers and patients, confirmed the need for eHealth/website delivery, and discussed potential topics of information. The illness representation or "Common Sense model of Self-Regulation" (CSM) focuses on how an individual's behaviour is influenced by his/her perceptions (40). Perceptions, in the case of the patient with an ICD, may be influenced by the reason for device implantation (41); short and long-term daily adaptations living with the device (42); receiving a shock (18); and the unpredictability of advanced heart failure (43). This model offers a sound theoretical framework to address the psychological and informational needs of patients with an ICD. Using the sixstage 'experience-based co-design' approach, professionals and service users worked in partnership (44-47) to select and optimize the composition of these components. Lessons learned from the development of a supportive intervention within the field of cancer care (48, 49) was implemented. The 'added' value of CHOICE-ICD is that it is a 'state-of-the-art' webbased intervention, made possible by an interdisciplinary team including software developers, patients and family members, with the patient remaining a central partner (50) in decisions. The finalized prototype of the intervention will now be pilot tested by patients within Northern Ireland and Glasgow, optimized based on feedback, before a clinical feasibility trial.

### 3: Aim & Objectives

An eHealth intervention co-designed by patients, family members and professionals will be feasible and acceptable, enabling progression to an effectiveness trial.

#### Aim of this study

Co-design and test an eHealth intervention for patients' pre-implantation and those recently implanted an ICD, together with family members and professionals.

### Objectives of this study

1. To co-develop and pilot test a prototype of an eHealth intervention with patients with an ICD, their family members and professionals.









- 2. To optimise and deliver the intervention to patients awaiting and those with an implanted ICD, with data collected to determine recruitment/demand, engagement with the intervention (System Usability Scale-SUS) & attrition.
- 3. To explore the acceptability of the intervention through a questionnaire and focus groups with patients, family members and healthcare professionals.
- 4. To undertake a process evaluation identifying methodological issues, face and psychometric validity and the primary outcome for a future trial. Self-reported data from validated questionnaires delivered pre- and post-intervention will measure patients' knowledge, attitudes and experiences (EOL-ICD), device acceptance and concerns (ICDc and Florida Patient Acceptance Survey), quality of life (EuroQol-5D), anxiety (BAI) and illness perceptions. Caregivers will complete the carer strain index (CSI)

### 4: Trial design:

This CHOICE-ICD methodology is framed according to the Medical Research Council (MRC) framework (36), and in accordance with the Common Sense model of Self-regulation and previous research conducted by the experienced research team (19, 27, 37, 51-54).

#### Methods:

This study comprises of two phases, outlined in the Consort diagram (Figure 1) (55) and Gantt chart (Appendix 1).

### Phase 1: Co-design the intervention (Objective 1)

The co-design of the intervention involved a number of iterative steps (48). Previous work conducted by this research team developed the concept of an eHealth intervention. The first integrated workshop stakeholders (n=18; patients with an ICD, family members, cardiologists, heart failure nurses, cardiac physiologists, and software developers) was held on the 8<sup>th</sup> September 2023. Interaction focused on balancing technical, holistic and practical details, with the provision of clinical facts without evoking fear, in order to create a patient-centred learning environment. Unstructured meetings (online) were held with 10 stakeholders (patient, family members and professionals) who tested and provided feedback on the prototype of the APP, which was conveyed at the forthcoming stakeholder meeting. The prototype was tested at each









iterative stage for two weeks. Within the second stakeholder workshop (n=16), on the 22nd May, feedback from testers (n=8) informed the components of the APP, including content, patient videos, VR option, ease of use and navigation. The intervention was further optimised and the testers, over a 2-week period, invited to provide feedback.

Field notes were recorded, with the discussion digitally recorded, transcribed verbatim and thematically analysed (LH). A consensus approach and agreement was sought on the development of the prototype of the intervention, in terms of content and presentation. Data analysis outlining the key components of the intervention was discussed and confirmed throughout, by the international advisory team. The web-based intervention was developed through an expert software developer- ProPeer solutions. This established company has successfully collaborated on a number of projects. Here are a few examples:- Treatment of patients suffering with Post Traumatic Stress Disorder <a href="https://youtu.be/6D5sNgjHtko">https://youtu.be/6D5sNgjHtko</a> Exercise Solution with Parkinson's

https://drive.google.com/file/d/1j5kPbDEJ95qK1RyHCuvKFVoXwewaLYF-/view?usp=sharing
\_The intervention was optimised through repeated discussions and agreement between research team, software developers and patients.

## Phase 2: Clinical study of the web-based intervention (Objectives 2-4)

Patients attending routine outpatient appointments at the Belfast Health and Social Care Trust (BHSCT) and Golden Jubilee National Hospital (GJNH), Clydebank will be identified and invited to participate by the Cardiologist or Heart Failure Nurse according to inclusion/exclusion criteria (See Table 1). The BHSCT and GJNH are busy tertiary centres, implanting collectively over 700 devices per annum (2019/2020). Written consent to pass on contact details to the researchers (LH or Research Assistant - RA) will be obtained. Patients will be asked to nominate a family member or caregiver, to participate in the study. Only when the patient has spoken to the family member/caregiver will their contact details be passed onto the researcher. Written information detailing the study will be provided and interested patients and family members will be offered one week to consider participation. The researcher (LH or RA) will make contact with the patient and family member to ensure both are agreeable to participate,









before obtaining written consent, baseline data is collected and 1:1 randomisation. Baseline questionnaires will be completed in all patients and caregivers recruited to the study. A convenience sample of *n*=64 patients will be randomised to the intervention and usual care, with n=64 receiving usual care alone, across Northern Ireland and Scotland. Patients and caregivers will be followed up at 3 months and 6 months' post intervention. Patients who received the Choice-ICD intervention, along with their caregivers and members of their clinical team (i.e heart failure nurse, cardiologist or cardiac physiologists) will be invited to participate in a focus group. Members of the clinical team (8-10) will be invited by the local collaborator (Dr Dixon or Prof Gardner) and if agreeable, contact details will be passed to the researcher to provide information on the study and obtain consent. Focus group will be conducted separately (Focus group 1: patients and caregivers Focus group 2: healthcare professionals) within each clinical site. Any patients, caregivers or healthcare professionals involved in Phase 1 (Codesign of the APP) will be excluded.

#### 5: Power calculations:

Unpublished audit data show that in 2019/2020: 482 ICD/CRTD were implanted in NI and 250 implanted in Scotland. Given the total population size of 732 patients, we need to recruit 128 patients in total to account for an expected 10% attrition rate. This would leave a sample size of n = 114 (intervention, n = 57; control, n = 57) that enables us to estimate a recruitment rate of 50% to within a 90% confidence interval of +/- 10%, which should provide an accurate representation of the patient population. These statistics have been deemed suitable as higher precision would warrant a larger sample size, with the required resources being unsuitable for a feasibility study. Co-applicant (MD) will provide statistical support throughout. The results of the proposed study will enable the planning of a future definitive trial.

Table 1: Eligibility Criteria

| Patient | Caregiver | Healthcare Professional |
|---|---|---|
| Patients with heart failure awaiting or with an ICD (no | Have contact with the patient at least 5 times per week. | |









| time restriction on implantation) | | defibrillator |
|---|---|---|
| Aged 18 years and over | Aged 18 and over. | Willing to provide written informed consent |
| No cognitive impairment | Be nominated by the patient. | Involved in the care of a patient using the Choice-ICD App |
| Willing to provide written informed consent | Be physically and mentally capable of participation (self-assessment) | |
| | Willing to provide written informed consent. | |

#### Exclusion criteria:

- Patients, judged by their Cardiologist as physically or mentally unsuitable to complete the study.
- · Patients or caregivers lacking capacity to give consent.
- Patients who have known pregnancy
- Caregivers who's patient is unwilling to take participate

#### 6: Intervention:

Patients and family members will receive the online intervention (accessed via a password protected link) and British Heart Foundation (BHF) booklet: "Implantable Cardioverter Defibrillators" (2018- HIS19/1117) or the BHF booklet only (usual care group). The eHealth intervention is theoretically driven, interactive and provides personalised information to patients and family members when and where they wish to access it. Topics include: "How does an ICD work? How will it affect my daily activities? What do I do if I experience a shock? Do I have choices ahead when my health declines?" Each topic will have a link to a printable fact sheet with a prompt card that patients can take with them to their next professional consultation. Five short (2-3 minutes) videos, involving patients, caregivers and professionals, developed with MacMillen Media, will be uploaded onto the APP, alongside animation clips and useful links to online resources (56). A discussion forum will be accessible for participants using the APP,









which will be closely moderated by the researcher, who will ensure any concerning posts or dialogue are promptly removed, and the necessary action is taken. The diary function will allow patients to record and be reminded of future appointments. This detail will not be collected, but rather is for the patient's use only. The intervention is both an informational support resource as well as a "prompt" for patients and professionals to engage in complex discussions. Patients and family members will engage with the intervention for 3 months.

Patients recruited from the Belfast Health and Social care Trust and randomised to receive the Choice -ICD intervention, will be invited to access the virtual reality (VR) enhanced intervention. Participants attending during their visit 1 or 2 to the BHSCT, will be invited to access the optional VR aspect. The VR enhanced intervention will be carried out within Queen's University premises at the time in which focus groups have been arranged. Interested patients will receive instructions on the use of the headset (Meta Quest 3) and supervised by the researcher while it is in place The session will last for a maximum of 10 minutes, therefore minimising risk of adverse effects. A protocol to ensure the safety and tolerability of the VR session has been developed. No data will be collected from the headset. Anonymised data linked to recruitment to the VR option will be collected.

#### 7: Data collection & Outcome Measures:

Descriptive data including recruitment/demand, participants' engagement/adherence with the intervention (*i.e.*, number of log-ins and screens viewed), and attrition will be collected, in line with the standards for feasibility studies (57). Patients will complete a paper copy of the validated patient reported outcome measures and short demographic questionnaire (*i.e.*, age, education, New York Heart Association (NYHA), and indication for device) at baseline. They will also complete paper versions of validated questionnaires, including the ICD concerns questionnaire (ICDC) (58), Experiences, Attitudes and Knowledge of End-of-Life issues in Implantable Cardioverter Defibrillator Questionnaire (EOL-ICDQ) (59), Beck Anxiety Inventory (BAI) (60), Brief Illness perception questionnaire (15), Florida Patient Acceptance Survey (FPAS) (61) and the Kansas City Cardiomyopathy questionnaire (KCCQ- 12) quality of life tool (62). Family members will complete the Carer Strain Index (CSI) (63). Questionnaires, at baseline, 3 and 6 months will be disseminated by the QUB researcher (LH) or research nurse









if the patient lives in Clydebank. Data will be collected month 3, including system usability scale, and again at month 6 (post intervention). Questionnaires will be disseminated in paper copy. At 3 and 6 months, a stamped addressed envelope will be provided to promote return of the questionnaires to the researcher at QUB (LH). Reasons regarding loss to follow-up will be monitored. <u>Primary outcome measures</u> are the feasibility, acceptability and usability (according to SUS) of the intervention. <u>Secondary outcome measures</u> are effect of the eHealth intervention on patients' knowledge, anxiety and device related quality of life as measured by the questionnaires. (Appendix 2)

All data collected will be monitored by the Chief Investigator to ensure ethical, legal or management issues arising are addressed promptly. The researcher (LH) alongside her team, have experience and publications in this area (LD, DF, MD, OS). Results from the study will be reported back to participants and inform the intervention in preparation for a larger future trial.

### 8: Data Analysis

Descriptive and inferential data analysis will be conducted by LH using SPSS (IDM Statistics 22), which will focus on calculating effect sizes that describe the differences between pre- and post-intervention. Sub-group analysis will be undertaken between patients implanted with an ICD for the first time and those with a pre-existing device. Qualitative data will be collected from two focus groups with patients and family members (n=20) at 3 months by the RA. Results will enrich understanding of the perceptions of patients and family members towards the intervention and its acceptability, the validated tools used and how the intervention may facilitate future deactivation conversations. Barriers and facilitators of the intervention will be openly discussed. A brief acceptability questionnaire will be completed (64). Two separate focus group with healthcare professionals (n=20) will enable an insight into their perspectives towards the intervention. Each focus group will be audio-recorded, transcribed verbatim and thematically analysed. The transcript will be independently analysed to improve rigour and consistency.

### 9: Trial Monitoring:









The study will also be monitored periodically by members of the International steering group, who will assess the progress of the study, verify adherence to the protocol and national requirements, and review the completeness, accuracy and consistency of the data.

International experts (Debra Moser, USA, Ingela Thylen, Sweden, Susanne Pedersen, Denmark), high volume device implanter and heart failure specialists (Nick McKeag, Kat McCreary) and cardiologists Stephen Pettit & Karen Hogg, two patient representatives from Patient support group and BHF representative will advise on all aspects of the study. Advice and support is also available from Dr Paul Best from the Centre of Technological Innovation, Mental health and Education (TIME).

The Research Governance Office at Queen's University Belfast, as lead sponsor, audits research studies conducted by University staff to make sure that they are being carried out in accordance with the Research Governance Framework and with the highest standards of integrity. Staff from the Research Governance Office may review the data collected in this study as part of their annual audit programme

#### 10: Trial Management:

The study will be managed by an expert team of researchers and clinicians. The researcher (LH) will be supervised by Prof Donna Fitzsimons, Prof Martin Dempster Dr Olinda Santin, Dr Lana Dixon and Prof Roy Gardner to ensure research integrity and that the project is completed on time. (Gantt chart- Appendix 1)

#### 11: Ethics

The protocol will be submitted to an NHS/HSC Research Ethics Commitee. Governance approval will be sought through the New HSC Approvals system <a href="New Research Approvals">New Research Approvals</a>
Service for HSC R&D in Northern Ireland | Public Health Agency - Research & Development in Northern Ireland (hscni.net) as well as approval within Golden Jubilee hospital, Clydebank and the Belfast HSC Trust. The Ethics Committees will be informed of all changes to the study









#### 12: Dissemination

The results will be published in peer review journal, as well presented at national and international congresses. Patients will have the opportunity to receive a copy of the results. Dissemination will also include regional meetings with patients and healthcare professionals.

#### 13: **References**

- 1. Connolly SJ, Hallstrom AP, Cappato R, Schron EB, Kuck KH, Zipes DP, et al. Meta-analysis of the implantable cardioverter defibrillator secondary prevention trials. AVID, CASH and CIDS studies. Antiarrhythmics vs Implantable Defibrillator study. Cardiac Arrest Study Hamburg. Canadian Implantable Defibrillator Study. Eur Heart J. 2000;21(24):2071-8--8.
- 2. Raatikainen MJP, Arnar DO, Zeppenfeld K, Merino JL. Statistics on the use of cardiac electronic devices and electrophysiological procedures in the European Society of Cardiology countries: 2014 report from the European Heart Rhythm Association. Europace. 2015;17:1-175.
- 3. Programme NCA. National Audit of Cardiac Rhythm management devices and ablation: 2016/2017 Summary Report London; 2019 11th July 2019.
- 4. Young JB, Abraham WT, Smith AL, Leon AR, Lieberman R, Wilkoff B, et al. Combined cardiac resynchronization and implantable cardioverter defibrillation in advanced chronic heart failure: the MIRACLE ICD Trial JAMA. 2003;289(20):2985-694.
- 5. McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Böhm M, et al. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021;42(36):3599-726.
- 6. Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Bloma N, Borggrefe M, Camm J, et al. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC. European Heart Journal. 2015;36:2793-867.
- 7. Nauffal V, Zhang Y, Tanawuttiwat T, Blasco-Colmenares E, Rickard J, Marine JE, et al. Clinical decision tool for CRT-P vs. CRT-D implantation: Findings from PROSE-ICD. Plos One. 2017;12(4):17520.
- 8. Saxon LA, Bristow MR, Boehmer J, Krueger S, Kass DA, De Marco T, et al. Predictors of sudden cardiac death and appropriate shock in the Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Trial. Circulation. 2006;114:2766-72.
- 9. Irvine J, Dorian P, Baker B, O'Brien BJ, Roberts R, Gent M, et al. Quality of life in the Canadian Implantable Defibrillator study (CIDS) AmHeart J. 2002;144:282-9.
- 10. Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, et al. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005;352(3):225-37.
- 11. Thylen I, Dekker RL, Jaarsma T, Stromberg A, Moser D. Characteristics associated with anxiety, depressive symptoms and quality of life in large cohort of Implantable Cardioverter Defibrillator recipients. J Psychosom Res. 2014;77:122-7.
- 12. Udlis KA. The Impact of Technology Dependency on Device Acceptance and Quality of Life in Persons with Implantable Cardioverter Defibrillators. Journal of Cardiovascular Nursing. 2013;28:E65-E73.
- 13. Wong FM, Sit JW, Wong EM, Choi KC. Factors associated with health-related quality of life among patients with implantable cardioverter defibrillator: identification of foci for nursing intervention. J Adv Nurs. 2014;70(12):2821-34.









- 14. Pedersen SS, van Domburg RT, Theuns DA, Jordaens L, Erdman RA. Type D personality is associated with increased anxiety and depressive symptoms in patients with an implantable cardioverter defibrillator and their partners. Psychosom Med. 2004;66(5):714-9.
- 15. Timmermans I, Versteeg H, Meine M, Pedersen SS, Denollet J. Illness perceptions in patients with heart failure and an implantable cardioverter defibrillator: Dimensional structure, validity, and correlates of the brief illness perception questionnaire in Dutch, French and German patients. J Psychosom Res. 2017;97:1-8.
- 16. Lewis KB, Stacey D, Matlock DD. Making decisions about Implantable Cardioverter- Defibrillators from implantation to end-of-life: an integrative review of patients' perspectives Patient. 2014;7:243-60.
- 17. Green AR, Jenkins A, Masoudi FA, Magid DJ, Kutner JS, Leff B, et al. Decision-Making Experiences of Patients with Implantable Cardioverter-Defibrillators. Pacing Clin Electrophysiol. 2016;39(10):1061-9.
- 18. Groarke J, Beirne A, Buckley U, O'Dwyer E, Sugrue D, Keelan T, et al. Deficiences in Patients' Comprehension of Implantable Cardioverter Defibrillator Therapy. PACE. 2012;35:1097.
- 19. Hill L, McIlfatrick S, Taylor BJ, Dixon L, Cole BR, Moser DK, et al. Implantable cardioverter defibrillator (ICD) deactivation discussions: Reality versus recommendations. Eur J Cardiovasc Nurs. 2016;15(1):20-9.
- 20. Pedersen SS, Knudsen C, Dilling K, Sandgaard NCF, Johansen JB. Living with an implantable cardioverter defibrillator: patients' preferences and needs for information provision and care options. Europace. 2017;19:983-90--90.
- 21. Lee MC, Sulmasy DP, Gallo J, Kub J, Hughes M, Russell S, et al. Decision-making of patients with implantable cardioverter-defibrillators at end-of-life. family members experience. American Journal of Hospice and Palliative Medicine. 2017;34(6).
- 22. Cowie MR, Anker SD, Cleland JGF, Felker GM, Filippatos G, Jaarsma T, et al. Improving care for patients with acute heart failure: before, during and after hospitalization. ESC Heart Fail. 2014;1(2):110-45.
- 23. McDonagh TA, Blue L, Clark AL, Dahlström U, Ekman I, Lainscak M, et al. European Society of Cardiology Heart Failure Association Standards for delivering heart failure care. Eur J Heart Fail. 2011;13:235-41--41.
- 24. Lampert R, Hayes DL, Annas GJ, Farley MA, Goldstein NE, Hamilton RM, et al. HRS consensus statement on the management of cardiovascular implantable electronic devices (CIEDs) in patients nearing end of life or requesting withdrawal of therapy. . Heart Rhythm. 2010;7:1008-26.
- 25. Padeletti L, Omar DO, Boncinelli L, Brachman J, Camm JA, Daubert JC, et al. EHRA expert consensus statement on the management of cardiovascular implantable electronic devices in patients nearing end of life or requesting withdrawal of therapy. . Europace. 2010;12:1480-9.
- 26. Hjelmfors L, Stromberg A, Friedrichsen M, Martensson J, Jaarsma T. Communicating prognosis and end of life care to heart failure patients: A survey of heart failure nurses' perspectives European Journal of Cardiovascular Nursing. 2014;13(2):152-61.
- 27. Hill L, McIlfatrick S, Taylor BJ, Jaarsma T, Moser D, Slater P, et al. Patient and Professional Factors That Impact the Perceived Likelihood and Confidence of Healthcare Professionals to Discuss Implantable Cardioverter Defibrillator Deactivation in Advanced Heart Failure: Results From an International Factorial Survey. J Cardiovasc Nurs. 2018;33(6):527-35.
- 28. Elwyn G, Laitner S, Coulter A, Walker E, Watson P, Thomson R. Implementing shared decision making in the NHS. BMJ. 2010;341:5146.
- 29. Ingadottir B, Thylén I, Jaarsma T. Knowledge expectations, self-care, and health complaints of heart failure patients scheduled for cardiac resynchronization therapy implantation. Patient Preference and Adherence. 2015;9:913-21.
- 30. Office National S. Internet users, UK: 2020. 2020.









- 31. Zippel-Schultz B, Palant A, Eurlings C, C FS, Hill L, Thompson DR, et al. Determinants of acceptance of patients with heart failure and their informal caregivers regarding an interactive decision-making system: a qualitative study. BMJ Open. 2021;11(6):e046160.
- 32. Schenker Y, Fernandez A, Sudore R, Schillinger D. Interventions to Improve Patient Comprehension in Informed Consent for Medical and Surgical Procedures: A Systematic Review. Medical Decision-making. 2011;31:151-73.
- 33. Barrett M, Boyne J, Brandts J, Brunner-La Rocca HP, De Maesschalck L, De Wit K, et al. Artificial intelligence supported patient self-care in chronic heart failure: a paradigm shift from reactive to predictive, preventive and personalised care. Epma j. 2019;10(4):445-64.
- 34. Ooi SL, He HG, Dong Y, Wang W. Perceptions and experiences of patients living with implantable cardioverter defibrillators: a systematic review and meta-synthesis. Health Qual Life Outcomes. 2016;14(1):160.
- 35. Pedersen SS, Skovbakke SJ, Wiil UK, Schmidt T, dePont Christensen R, Brandt CJ, et al. Effectiveness of a comprehensive interactive eHealth intervention on patient-reported and clinical outcomes in patients with an implantable cardioverter defibrillator [ACQUIRE-ICD trial]: study protocol of a national Danish randomised controlled trial. BMC Cardiovasc Disord. 2018;18(1):136.
- 36. Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Bmj. 2008;337:a1655.
- 37. Hill L, McIlfatrick S, Taylor B, Dixon L, Harbinson M, Fitzsimons D. Patients' perception of implantable cardioverter defibrillator deactivation at the end of life 2014; <a href="http://pmj.sagepub.com/content/early/2014/09/17/0269216314550374(Journal, Electronic)">http://pmj.sagepub.com/content/early/2014/09/17/0269216314550374(Journal, Electronic)</a>.
- 38. Hill LM, McIlfatrick S, Taylor B, Dixon L, Fitzsimons D. Implantable cardioverter defibrillator (ICD) functionality: patient and family information for advanced decision-making. BMJ Support Palliat Care. 2019.
- 39. Millerick Y. British Heart Foundation heart failure palliative care project report: The Glasgow and Clyde experience. London: British Heart Foundation; 2010.
- 40. Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016;39(6):935-46.
- 41. Rahmawati A, Chishaki A, Ohkusa T, Sawatari H, Tsuchihashi-Makaya M, Ohtsuka Y, et al. Influence of primary and secondary prevention indications on anxiety about the implantable cardioverter-defibrillator. J Arrhythm. 2016;32(2):102-7--7.
- 42. Flemme I, Johansson I, Strömberg A. Living with life-saving technology coping strategies in implantable cardioverter defibrillators recipients. J Clin Nurs. 2012;21(3-4):311-21.
- 43. Hill L, Prager Geller T, Baruah R, Beattie JM, Boyne J, de Stoutz N, et al. Integration of a palliative approach into heart failure care: a European Society of Cardiology Heart Failure Association position paper. Eur J Heart Fail. 2020.
- 44. Aidemark J, Askenäs, L., Nygårdh, A., Strömberg, A. . User Involvement in the Co-design of Self-care Support Systems for Heart Failure Patients. Procedia computer science. 2015;64:118-24.
- 45. Fund. TK. Experience-based co-design. Working with patients to improve healthcare 2019 [Available from: <a href="http://www.kingsfund.org.uk/projects/ebcd">http://www.kingsfund.org.uk/projects/ebcd</a>.
- 46. Paton N, Callander R, Cavill M, et al. Collaborative quality improvement: consumers, carers and mental health service providers working together in service co-design. Australas Psychiatry. 2013;21(1):78-9--9.
- 47. O'Brien N, Heaven B, Teal G, et al. Integrating evidence from systematic reviews, qualitative reserach and expert knowledge using co-design techniques to develop a web-based intervention for patients in the retirement transition. Journal of Medical Internet Research. 2016;18(8).









- 48. Santin O, McShane T, Hudson P, Prue G. Using a six-step co-design model to develop and test a peer-led web-based resource to support informal carers of cancer patients. Psycho-oncology. 2019;28(3):518-24--24.
- 49. Tsianakas V, Robert G, Maben J, et al. Implementing patient-centred cancer care: using experience-based co-design to improve patient experience in breast and lung cancer services. Support Care Cancer. 2012;20(11):2639-47--47.
- 50. Ekman I, Wolf A, Olsson L, Taft C, Dudas K, Schaufelberger M, et al. Effects of person-centred care in patients with chronic heart failure: the PCC-HF study. European Heart Journal. 2012;33:1112-9.
- 51. Doherty LC, Fitzsimons D, McIlfatrick SJ. Carers' needs in advanced heart failure: A systematic narrative review. Eur J Cardiovasc Nurs. 2016;15(4):203-12.
- 52. Dempster M, Howell D, McCorry NK. Illness perceptions and coping in physical health conditions: A meta-analysis. J Psychosom Res. 2015;79(6):506-13.
- 53. Perera SM, O'Callaghan C, Ugalde A, Santin O, Beer C, Prue G, et al. Codesigning a supportive online resource for Australian cancer carers: a thematic analysis of informal carers' and healthcare professionals' perspectives about carers' responsibilities and content needs. BMJ Open. 2021;11(10):e055026.
- 54. Santin O, Jenkins C, Nghiem HLP, Prue G, Reid J, Lohfeld L, et al. The development of a web-based resource to provide information and psychosocial support to informal cancer carers in hospitals in Vietnam. Psychooncology. 2020;29(5):920-6.
- 55. Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, et al. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot and Feasibility Studies. 2016;2:64-.
- 56. The heart teams' role in ICD management throughout the life course: clinical and ethical challenges. ESC Congress; 2016; Rome: European Society of Cardiology.
- 57. Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, et al. How we design feasibility studies. Am J Prev Med. 2009;36(5):452-7.
- 58. Frizelle DJ, Lewin B, Kaye G, Moniz-Cook ED. Development of a measure of the concerns held by people with implanted cardioverter defibrillators: The ICDC. British Journal of Health Psychology. 2006;11:293-301-293-301.
- 59. Thylen I, Wenemark M, Fluur C, Stromberg A, Bolse K, Arestedt K. Development and evaluation of the EOL-ICDQ as a means of experiences, attitudes and knowledge in end-of-life in patients living with an implantable cardioverter defibrillator. European Journal of Cardiovascular Nursing. 2014;13(2):142-51.
- 60. Berg SK, Rasmussen TB, Herning M, Svendsen JH, Christensen AV, Thygesen LC. Cognitive behavioural therapy significantly reduces anxiety in patients with implanted cardioverter defibrillator compared with usual care: Findings from the Screen-ICD randomised controlled trial 2019; (Journal, Electronic):[24th October 2019-doi: 10.1177/2047487319874147 pp.].
- 61. Burns JL, Serber ER, Keim S, Sears SF. Measuring patient acceptance of implantable cardiac device therapy: initial psychometric investigation of the Florida Patient Acceptance Survey. J Cardiovasc Electrophysiol. 2005;16(4):384-90.
- 62. Spertus JA, Jones PG. Development and Validation of a Short Version of the Kansas City Cardiomyopathy Questionnaire. *Circ Cardiovasc Qual Outcomes*. 2015;8:469-476.
- 63. Robinson B. Validation of a Caregiver Strain Index. Journal of Geriat Soc. 1983;38:344-8--8.
- 64. Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, et al. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017;12(1):108.









## 14: Appendices

### Appendix 1: Gantt chart of the project











# Appendix 2:

Feasibility outcomes & Progression rules: description and target

| Measure | Description of outcome | Target: a priori<br>Criteria for<br>success |
|---|---|---|
| Recruitment Rate | Proportion of eligible participants identified who participated in the study | 60% |
| Completion of data collection measures (baseline, 3 & 6 months) | Proportion of consented participants who completed all questionnaires at baseline and post-intervention | 60% |
| Patient engagement | Proportion of participants who completed all topics | 60% |
| Participant acceptability | Proportion of patients accessing the intervention found it clear and understandable | 80% |
| Intervention acceptability | Proportion of patients, caregivers and professionals who accessed the intervention and would use it again | 80% |

If the number is within 5% points of the progression target, a discussion would occur regarding progression to future trial within the research team